CLINICAL TRIAL: NCT06977750
Title: A Multicenter, Randomized, Double-blind, Positive Controlled Clinical Study on the Efficacy and Safety of Succinylated Gelatin Electrolyte Sodium Acetate Injection for Acute Isovolumetric Hemodilution (ANH) in Elective Surgery
Brief Title: Clinical Study on the Effectiveness and Safety of Succinylated Gelatin Electrolyte Sodium Acetate Injection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPXMJDJZ-III01
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Normovolemic Hemodilution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental grou (Experimental)
  Interventions: Drug: succinylated gelatin electrolyte sodium acetate injection
- control group (Active Comparator)
  Interventions: Drug: succinylated gelatin electrolyte sodium acetate injection 1

INTERVENTIONS:
Drug: succinylated gelatin electrolyte sodium acetate injection 1 — Nanjing Chia-Tai Tianqing Pharmaceutical Company
  Arms: control group
Drug: succinylated gelatin electrolyte sodium acetate injection — Gelaspan
  Arms: experimental grou

SUMMARY:
The succinylated gelatin electrolyte sodium acetate injection (specification: 500 mL: 20 g) developed and produced by Nanjing Chia-tai Tianqing Pharmaceutical. is used as the experimental drug, and the succinylated gelatin electrolyte sodium acetate injection (trade name: Jialeban) produced and licensed by Braun Medical (Suzhou) Co., Ltd ®； Specification: 500 mL: 20 g) is used as a control drug to evaluate the clinical equivalence of two formulations in patients planning elective surgery by comparing the changes in stroke volume (SV) between 5 minutes after completion of ANH and immediately before the start of ANH.

ELIGIBILITY:
Inclusion Criteria:

1. Age range is 18 to 65 years old (including boundary values), with no gender restrictions.
2. Weight not less than 50 kg, weight not more than 100 kg, body mass index [BMI=weight (kg)/height 2 (m2)] within the range of 19.0~30.0 kg/m2 (including critical values).
3. Planned elective surgery with an estimated duration of less than 6 hours.
4. The expected ANH blood collection volume is 10% to 15% of the total blood volume.
5. Prior to enrollment, the Hb level of the subjects was ≥ 110 g/L.
6. The American Society of Anesthesiologists (ASA) has a rating of I-III.
7. Voluntarily participate in this experiment and sign a written informed consent form.

Exclusion Criteria:

1. Individuals with a history of severe cerebrovascular disease or severe mental illness, who have been deemed unsuitable by the researchers to participate in this trial.
2. Previous indications include heart valve disease, aortic stenosis, and severe peripheral vascular disease (such as a history of arteriosclerosis), and the researchers have determined that they are not suitable to participate in this trial.
3. Suffering from serious heart diseases, including but not limited to unstable angina, cerebrovascular accidents or transient ischemic stroke (within 6 months before screening), myocardial infarction (within 6 months before screening), New York Heart Association (NYHA) classification ≥ III, congestive heart failure, severe arrhythmia with poor drug control, requiring mechanical maintenance (such as pacemakers), placing heart stents or abnormal results of echocardiography and/or 12 lead electrocardiogram during screening, has clinical significance.
4. Patients with hypertension have poor blood pressure control (SBP ≥ 160mmHg and/or DBP ≥ 100mmHg), and cannot discontinue long-term antihypertensive drugs such as angiotensin-converting enzyme inhibitors/angiotensin II receptor antagonists and potassium sparing diuretics 10 hours before surgery, and the researchers have determined that they are not suitable to participate in this trial.
5. Individuals with a history of liver cirrhosis or liver dysfunction during screening and deemed unsuitable for surgery by researchers: AST or ALT>2 times the upper limit of normal values; Albumin level<35 g/L; Blood bilirubin is greater than 1.5 times the upper limit of normal value.
6. Patients with abnormal renal function assessment during screening and deemed unsuitable for surgery by researchers: Cr or BUN>1.5 times the upper limit of normal values.
7. There are any of the following respiratory management risks during screening: 1) history of asthma (such as allergic asthma), wheezing; 2) Individuals with sleep apnea syndrome;
8. Hematological disorders such as sickle cell anemia, thalassemia, and pheochromocytoma.
9. There is a significant risk of bleeding or coagulation disorders, and the researchers assess that surgery is not suitable, including but not limited to: a) past/current thrombotic or thromboembolic events, or an increased risk of thrombotic or thromboembolic events; b) Require the use of antiplatelet or anticoagulant drugs (such as warfarin and clopidogrel) other than aspirin (up to 100 mg/d); c) Having a history of gastrointestinal, intracerebral hemorrhage, or other events considered severe bleeding, such as bleeding caused by the use of nonsteroidal anti-inflammatory drugs; d) PT prolongation>upper limit of normal value of 3 seconds or APTT prolongation>upper limit of normal value of 10 seconds, and the researcher evaluates it as unsuitable for surgery; e) PLT<80 × 109/L.
10. Diabetes patients with poor control, such as glycosylated hemoglobin ≥ 7%, and the investigator judged that they were not suitable to participate in the trial.
11. History of malignant tumors (excluding non metastatic basal cell carcinoma or squamous cell carcinoma, papillary thyroid carcinoma, and cervical cancer in situ that have been cured for ≥ 5 years and do not require follow-up).
12. Excessive blood volume (such as polycythemia vera) and fluid overload (such as systemic edema).
13. There is an active infection with poor control, which the researchers believe makes the subjects unsuitable to participate in this clinical study.
14. Preoperative complications include pulmonary edema, dehydration, burns, intestinal obstruction, critical illnesses such as sepsis, multiple organ failure, respiratory distress syndrome, organ transplantation, shock, etc.
15. When screening, there is a water electrolyte imbalance (such as hypercalcemia, hyperkalemia, etc.) and the researcher believes that the abnormality has clinical significance and is not suitable to participate in this clinical study.
16. Having undergone major surgeries or surgical incisions that have not fully healed within the first 6 months of screening: Major surgeries include but are not limited to any surgeries with significant bleeding risks, prolonged general anesthesia periods, or significant traumatic injuries.
17. Received anemia related treatment, colloidal solution, and/or blood products 14 days before surgery.
18. Those who have received the vaccine within one month before surgery.
19. Individuals who are known to be allergic to any component of the investigational drug; Known to be allergic to meat, especially red meat (mammalian meat) or internal organs; Known individuals who are allergic to lactose - α -1,3-galactose; And subjects with a history of severe allergic reactions (such as urticaria, angioedema, etc.).
20. Has a history of drug abuse in the past.
21. Patients who cannot discontinue corticosteroids, nonsteroidal anti-inflammatory drugs, cyclosporine, tacrolimus, or succinylcholinergic drugs within 7 days before surgery (or within 5 half lives of the drug, whichever is shorter).
22. Pregnant or lactating women, as well as male subjects (or their partners) or female subjects who have a pregnancy plan or are unwilling to use at least one medically recognized effective contraceptive measure (such as intrauterine device or condom) during the study period until 1 month after the last use of medication.
23. Those who have participated in any other non observational clinical trials and used the study drug or device within one month prior to the trial;
24. Participants may not be able to complete this study due to other reasons or may have other reasons deemed inappropriate by the researchers to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in stroke volume (SV) 5 minutes after completion of ANH compared to immediately before the start of ANH | 5 minutes after the completion of ANH compared to immediately before the start of ANH

CONTACTS AND LOCATIONS:
Overall Officials: wen ouyang, Principal Investigator — The Third Xiangya Hospital of Central South University; saiying wang, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- Third Xiangya Hospital of Central South University, Changsha, Hunan, China